CLINICAL TRIAL: NCT05889559
Title: Evaluation of the Diagnostic and Therapeutic Value of Tissue Ultrafiltration in Patients at Risk of Acute Compartment Syndrome (ACS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00268346
Record Dates: First submitted 2023-04-17; First posted 2023-06-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Acute Compartment Syndrome; Fracture, Bone; Tibial Fractures
MeSH Terms: conditions — Fractures, Bone; Tibial Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Pressure Monitoring Group (No Intervention): Participants in this group will have pressure monitoring of the anterior compartment of their leg using an indwelling IMP catheter (MY01, MY01 Inc., Montreal, CA). The participants will be treated according to the standard-of-care regarding management of their underlying injury and diagnosis of ACS as practiced by their treating surgeon. Participants will be followed for six months post-injury.
- Tissue Ultrafiltration Intervention Group (TUF) (Experimental): Participants in this group will have pressure monitoring of the anterior compartment of their leg using an indwelling IMP catheter (MY01, MY01 Inc., Montreal, CA). The participants will be treated according to the standard-of-care regarding management of their underlying injury and diagnosis of ACS as practiced by their treating surgeon. In addition, participants in this group will will undergo three TUF of the anterior compartment of the injured limb. Participants will be followed for six months post-injury.
  Interventions: Device: Tissue Ultrafiltration Catheters

INTERVENTIONS:
Device: Tissue Ultrafiltration Catheters — patients randomized to the experimental arm will have three TUF catheters placed in the anterior muscle compartment of the injured limb. The TUF catheters will be connected to a closed suction drain and will remove interstitial fluid from the muscle.
  Arms: Tissue Ultrafiltration Intervention Group (TUF)

SUMMARY:
The goal of this clinical trial is to learn if tissue ultrafiltration (TUF) catheters can reduce intramuscular pressure and prevent acute compartment syndrome (ACS) in adults ages 18-60 with severe proximal tibia or tibial shaft fractures.

The main questions it aims to answer are:

Will intramuscular pressure (IMP) be lower in the TUF cohort compared to controls?

Will the consensus likelihood of ACS, incidence of fasciotomy, and 6-month functional outcomes be better in the TUF cohort?

Are interstitial fluid biomarkers predictive of ACS?

Researchers will compare patients randomized to TUF catheters (n=30) versus control patients receiving standard-of-care only (n=30) to see if TUF lowers ACS risk and improves recovery.

Participants will:

Be enrolled within 14 hours of injury or prior to high-risk surgery within 48 hours.

Receive continuous anterior compartment pressure monitoring.

Undergo standard-of-care clinical evaluation and treatment.

(TUF arm only) Have three TUF catheters placed in the injured limb to remove interstitial fluid.

Return for a 6-month follow-up to assess complications, healing, muscle function, and patient-reported outcomes.

(Hennepin Healthcare subset) Provide interstitial fluid samples for biomarker analysis.

DETAILED DESCRIPTION:
The study will enroll 60 adults ages 18-60 admitted to the hospital with severe open or closed fractures of the proximal tibia or tibial shaft at risk for ACS. Participants will be randomized to either treatment with tissue ultrafiltration (TUF) catheters (n=30) or to a control group (n=30). Patients will be enrolled within 14 hours of initial injury, or just prior to undergoing surgical procedures that are associated with a risk of post-operative ACS within 48 hours of injury. All patients will receive continuous pressure monitoring of the anterior compartment of their leg. Both groups will receive comprehensive clinical evaluation and will be treated according to the standard-of-care regarding management of their underlying injury and diagnosis of ACS as practiced by their treating surgeon. In addition, patients randomized to the experimental arm will have three TUF catheters placed in the anterior muscle compartment of the injured limb. The TUF catheters will be connected to a closed suction drain and will remove interstitial fluid from the muscle. All patients will be followed at 6 months following initial hospital discharge. This visit will include a clinical evaluation of complications, hospital admission and emergency room visits, wound and fracture healing, infection, muscle sensory and function exam and patient-reported outcome.

We hypothesize that intramuscular pressure (IMP) will be lower in the TUF cohort compared to controls. In addition, we expect that the expert panel consensus likelihood of ACS, defined as the median of the ratings of the individual panel members who evaluated each patient, and the incidence of fasciotomy will be lower in the TUF cohort. Finally, patients in the TUF cohort will demonstrate superior functional outcome at 6 months following injury compared to those in the control cohort, levels of specific biomarkers as measured in the interstitial fluid will be worse in patients with ACS compared to patients without ACS in the treatment group, and there will be a threshold for each biomarker which is predictive of ACS (biomarkers will be collected from at least 10 patients/ up to full sample of intervention arm patients enrolled at Hennepin Healthcare only).

ELIGIBILITY:
INCLUSION CRITERIA The target population for this study include adults ages 18-60 with high-energy injuries of the upper leg considered at risk for ACS at time of admission by virtue of their mechanism of injury, fracture pattern, clinical signs, or need to undergo fracture fixation surgery (internal or external fixation) within 48 hours of admission. Recruitment of participants will happen during hospital admission for treatment of injury.

Eligible patients must meet all of the following criteria and be enrolled during one of two possible times: within 14 hours of injury, or prior to undergoing surgical intervention (internal or external fixation on the injured limb) within 48 hours of admission. Eligible patients will be:

1. Between the ages of 18 and 60 years
2. Have sustained a high-energy upper leg injury such as open or closed proximal tibial shaft fracture with displacement, comminution, or segmental pattern; proximal fibula fracture; bicondylar tibial plateau fracture; Schatzker IV medial knee fracture-dislocation; proximal leg injury due to shotgun, rifle, or other projectile, or severe crushing injury.
3. Patient can be enrolled in the study and study procedures initiated within 14 hours of injury,* or be enrolled prior to undergoing urgent surgical intervention on the injured limb (defined as internal or external fixation) within 48 hours of admission.
4. Patient (or authorized legal representative) willing to sign informed consent.

   * If a patient has an eligible injury and is going to surgery within 2 hours (except for fasciotomy - which is an exclusion criteria), the patient can be enrolled and the study procedures initiated at the end of surgery. If an eligible patient is enrolled and there is no surgery anticipated within 2 hours, initiate study procedures immediately.

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patients not willing to participate
2. Patients with non-traumatic cases of acute compartment syndrome (e.g. severe exertion, snakebite, high-pressure injection injury)
3. Patients diagnosed with ACS or impending ACS such that immediate fasciotomy is recommended
4. Soft tissue wounds, including lacerations or abrasions, that are in a location that will interfere with safe insertion of indwelling pressure or TUF catheters (anterior - anterolateral aspect of the leg)
5. Patients not likely to follow-up (are homeless, incarcerated, live out-of-state).
6. Patients with known peripheral vascular disease
7. Non-ambulatory due to an associated complete spinal cord injury; Non-ambulatory before the injury due to a pre-existing condition.
8. Very low clinical concern for ACS at time of admission.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To test whether TUF reduces Intramuscular Pressure (IMP) compared to control patients. | 6 months post injury
  Proportion of patients with a of Change in continuously measured IMP.

SECONDARY OUTCOMES:
To test whether there are differences in the incidence of ACS in patients with severe leg injuries treated with active TUF compared to the control group. | 6 months post injury
  The consensus likelihood of ACS as assessed by a panel of experts after review of a standardized patient profile.
To test whether TUF reduces the incidence of fasciotomy compared to control patients. | 6 months post injury
  Proportion of patients with a fasciotomy.
To test the impact of TUF on improving patient Global Health | 6 months post injury
  Veteran Rand 12 Health Survey (VR12)
To test the impact of TUF on improving patient physical function | 6 months post injury
  PROMIS Physical Function

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland School of Medicine R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - Atrium Health Musculoskeletal Institute, Charlotte, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee